CLINICAL TRIAL: NCT00002760
Title: A PHASE III TWO-ARM RANDOMIZED STUDY COMPARING ANTIANDROGEN WITHDRAWAL ALONE VERSUS ANTIANDROGEN WITHDRAWAL COMBINED WITH KETOCONAZOLE AND HYDROCORTISON IN PATIENTS WITH ADVANCED PROSTAGE CANCER
Brief Title: Antiandrogen Withdrawal in Treating Patients With Hormone-Refractory Prostate Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CALGB-9583; U10CA031946 (NIH); CLB-9583; CDR0000064708 (Registry Identifier: NCI Physician Data Query)
Record Dates: First submitted 1999-11-01; First posted 2004-07-19 (Estimated); Last update posted 2016-06-28 (Estimated); Status verified 2016-06

CONDITIONS: Prostate Cancer
Keywords: adenocarcinoma of the prostate; recurrent prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Ketoconazole; Hydrocortisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Antiandrogen withdrawal (Other): antiandrogen therapy withdrawn; patient who progress will be "crossed over" to Arm 1A: 400 mg ketoconazole PO tid and hydrocortisone 30 mgs PO q am and 10 mgs PO qhs until treatment is no longer effective
  Interventions: Other: Withdrawal of antiandrogen therapy
- Antiandrogen withdrawal + therapy (Active Comparator): Ketoconazole and hydrocortisone
  Interventions: Drug: ketoconazole; Drug: therapeutic hydrocortisone

INTERVENTIONS:
Drug: ketoconazole — 400 mg PO tid for as long as treatment is effective
  Arms: Antiandrogen withdrawal + therapy
Drug: therapeutic hydrocortisone — hydrocortisone 30 mg PO q am and 10 mg PO qhs for as long as treatment is effective
  Arms: Antiandrogen withdrawal + therapy
Other: Withdrawal of antiandrogen therapy — no drugs given
  Arms: Antiandrogen withdrawal

SUMMARY:
RATIONALE: Antiandrogen withdrawal may be an effective treatment for prostate cancer.

PURPOSE: Randomized phase III trial to study the effectiveness of ketoconazole and hydrocortisone for antiandrogen withdrawal in treating men with prostate cancer that is refractory to hormone therapy.

DETAILED DESCRIPTION:
OBJECTIVES: I. Compare the response rate and duration of response to antiandrogen withdrawal alone vs. antiandrogen withdrawal plus ketoconazole/hydrocortisone in patients with advanced hormone-refractory prostate cancer. II. Compare the response rate and duration of response to ketoconazole/hydrocortisone in patients treated with previous vs. simultaneous antiandrogen withdrawal. III. Evaluate the proportion of patients with circulating prostate cancer cells identified by reverse transcriptase-polymerase chain reaction (rt-PCR). IV. Determine whether rt-PCR positively correlates with response. V. Compare the likelihood of response to these regimens in patients whose prior hormonal therapy consisted of initial combined androgen blockage vs. initial monotherapy followed later by an antiandrogen. VI. Correlate adrenal androgen synthesis suppression, as measured by levels of various adrenal androgens, with response.

OUTLINE: Randomized study. Patients who develop progressive disease on Arm I cross to Arm II. Arm I: Antiandrogen Withdrawal. Antiandrogen stopped. Arm II: Antiandrogen Withdrawal plus Adrenal Androgen Blockade. Antiandrogen stopped; plus Ketoconazole, KCZ; Hydrocortisone, HC, NSC-10483.

PROJECTED ACCRUAL: Approximately 250 patients will be entered over 3 years to attain 238 eligible patients (including 25-40 minority patients).

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically diagnosed adenocarcinoma of the prostate Progressive metastatic or regional nodal disease after at least 4 weeks on flutamide, bicalutamide, or nilutamide, i.e.: Greater than 25% increase in sum of products of perpendicular diameters of all measurable lesions not previously irradiated OR Prostate-specific antigen (PSA) at least 5 ng/mL and risen from baseline on at least 2 successive occasions at least 2 weeks apart PSA progression required for "bone only" disease or disease that responded to androgen deprivation and is negative on imaging scans at entry Primary testicular androgen suppression with a luteinizing hormone-releasing hormone (LHRH) analogue plus antiandrogen or by orchiectomy required Intermittent LHRH analog/antiandrogen therapy resumed at least 4 weeks prior to and continued at time of entry LHRH analogue continued throughout study in absence of orchiectomy

PATIENT CHARACTERISTICS: Age: Any age Performance status: 0-2 Hematopoietic: Not specified Hepatic: Bilirubin no greater than 1.5 times normal AST no greater than 3 times normal Renal: Not specified Other: No active, uncontrolled condition including: Bacterial, viral, or fungal infection Hyperglycemia Gastric or duodenal ulcer No existing medical condition requiring systemic corticosteroids (inhaled and topical steroids allowed) No concurrent use of the following: Terfenadine Astemizole Cisapride

PRIOR CONCURRENT THERAPY: No prior therapy with experimental agents for metastatic disease Biologic therapy: No prior immunotherapy for metastatic disease Chemotherapy: No prior estramustine or other chemotherapy for metastatic disease Endocrine therapy: See Disease Characteristics No prior hormonal therapy for metastatic disease No prior aminoglutethimide No prior ketoconazole No prior hydrocortisone or other corticosteroids Prior experimental hormonal therapy requires approval of study chair Radiotherapy: At least 4 weeks since radiotherapy (8 weeks since strontium therapy) Surgery: Orchiectomy allowed

Max Age: 120 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 260 (Actual)
Dates: Start 1996-08; Primary Completion 2004-03 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Response: PSA | q 8 wks, at cross over (if applicable), at progression; q 6 mon in f/u

SECONDARY OUTCOMES:
Circulating prostate cancer cells | Pre treatment, 1 time
  Circulating prostate cancer cells as detected by rt-PCR will be correlated with outcomes
Adrenal androgen synthesis suppression | pre tx, after 1 and 3 months tx, at progression
  Adrenal androgen synthesis suppression will be assessed vs response

CONTACTS AND LOCATIONS:
Overall Officials: Eric Small, MD, Study Chair — University of California, San Francisco
Locations (2):
- United States (2):
  - UCSF Cancer Center and Cancer Research Institute, San Francisco, California
  - University of Minnesota Cancer Center, Minneapolis, Minnesota

REFERENCES:
- [Background] D'Amico AV, Halabi S, Vogelzang NJ, et al.: A reduction in the rate of PSA rise following chemotherapy in patients with metastatic hormone refractory prostate cancer (HRPC) predicts survival: results of a pooled analysis of CALGB HRPC trials. [Abstract] J Clin Oncol 22 (Suppl 14): A-4506, 383s, 2004.
- [Background] Halabi S, Small EJ, Kantoff PW, Kattan MW, Kaplan EB, Dawson NA, Levine EG, Blumenstein BA, Vogelzang NJ. Prognostic model for predicting survival in men with hormone-refractory metastatic prostate cancer. J Clin Oncol. 2003 Apr 1;21(7):1232-7. doi: 10.1200/JCO.2003.06.100. PMID 12663709
- [Background] Gilligan TD, Halabi S, Kantoff PW, et al.: African-American race is associated with longer survival in patients with metastatic hormone-refractory prostate cancer (HRCaP) in four randomized phase III Cancer and Leukemia Group B (CALGB) trials. [Abstract] Proceedings of the American Society of Clinical Oncology 21: A-725, 2002.
- [Result] Ryan CJ, Halabi S, Ou SS, Vogelzang NJ, Kantoff P, Small EJ. Adrenal androgen levels as predictors of outcome in prostate cancer patients treated with ketoconazole plus antiandrogen withdrawal: results from a cancer and leukemia group B study. Clin Cancer Res. 2007 Apr 1;13(7):2030-7. doi: 10.1158/1078-0432.CCR-06-2344. PMID 17404083
- [Result] Ryan CJ, Halabi S, Kaplan E, et al.: Use of adrenal androgen levels to predict response to ketoconazole in patients with androgen independent prostate cancer: results from CALGB 9583. [Abstract] J Clin Oncol 22 (Suppl 14): A-4558, 396s, 2004.
- [Result] Small EJ, Halabi S, Dawson NA, Stadler WM, Rini BI, Picus J, Gable P, Torti FM, Kaplan E, Vogelzang NJ. Antiandrogen withdrawal alone or in combination with ketoconazole in androgen-independent prostate cancer patients: a phase III trial (CALGB 9583). J Clin Oncol. 2004 Mar 15;22(6):1025-33. doi: 10.1200/JCO.2004.06.037. PMID 15020604
- [Result] Halabi S, Small EJ, Hayes DF, Vogelzang NJ, Kantoff PW. Prognostic significance of reverse transcriptase polymerase chain reaction for prostate-specific antigen in metastatic prostate cancer: a nested study within CALGB 9583. J Clin Oncol. 2003 Feb 1;21(3):490-5. doi: 10.1200/JCO.2003.04.104. PMID 12560440
- [Result] Halabi S, Small E, Farmer D, et al.: Reverse transcriptase polymerase chain reaction (RT-PCR) for prostate specific antigen (PSA) as a prognostic factor for survival among androgen independent prostate cancer patients (AICaP): a companion study to CALGB 9583. [Abstract] Proceedings of the American Society of Clinical Oncology 20: A-700, 2001.
- [Result] Vogelzang NV, Halabi S, Picus J, et al.: Prospective assessment of adrenal androgen levels as predictors of survival in androgen independent prostate cancer patients treated with ketoconazole: a correlative study to CALGB protocol 9583. [Abstract] Proceedings of the American Society of Clinical Oncology 20: A-749, 2001.